CLINICAL TRIAL: NCT00996957
Title: A Phase 1 Open-Label, Multiple Dose, Dose Escalation Study of ACE-041 in Patients With Advanced Solid Tumors or Relapsed/Refractory Multiple Myeloma
Brief Title: Study of ACE-041 in Patients With Advanced Solid Tumors or Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A041-01; dalantercept (Other: USAN)
Record Dates: First submitted 2009-10-09; First posted 2009-10-16 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Advanced Solid Tumors; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ALK1-Fc fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACE-041 (Experimental): Patients assigned to 1 of 9 possible dosing groups
  Interventions: Biological: ACE-041

INTERVENTIONS:
Biological: ACE-041 — Subcutaneous dose of ACE-041 approximately once every 3 weeks for a total of 4 doses. If disease stays the same or gets better, additional study drug may be offered.

SUMMARY:
For cancer cells to grow, they need to have nutrients supplied to them through blood vessels. The study drug, ACE-041, is designed to work by blocking the growth of those blood vessels and preventing cancer cells from growing. The purpose of this study is to establish safe dose levels of ACE-041 in patients with advanced solid tumors or relapsed/refractory multiple myeloma following multiple dose administration. This study will also evaluate if ACE-041 has an effect on tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic or unresectable advanced solid tumors (solid tumors must be measurable) or relapsed/refractory multiple myeloma for which the disease has progressed despite available standard therapies or for which no standard therapy exists.
* Life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0, 1, or 2 (not declining within 2 weeks prior to study day 1).

Exclusion Criteria:

* Central nervous system (CNS) metastases.
* Chemotherapy or other anti-cancer therapy within 4 weeks prior to study day 1, and/or nitrosoureas within the 6 weeks prior to study day 1.
* Lack of recovery from all toxic effects of previous chemotherapy, radiation therapy, biologic therapy, and/or experimental therapy with the exception of alopecia.
* Radiation therapy within 4 weeks prior to study day 1.
* Clinically significant pulmonary, cardiovascular, endocrine, neurologic, gastrointestinal or genitourinary disease unrelated to underlying solid tumor or multiple myeloma
* Significant cardiac risk (e.g. history of myocardial infarction, unstable angina, pulmonary hypertension, clinically significant arrhythmia, congestive heart failure within 1 year prior to study day 1).
* Diagnosis or family history of hereditary hemorrhagic telangiectasia.
* Major surgery within 6 weeks prior to study day 1.
* Parenteral antibiotics, or any life-threatening or active infection requiring parenteral antibiotic therapy within 1 month prior to study day 1.
* Therapeutic anti-coagulation.
* Uncontrolled hypertension.
* Autoimmune or hereditary hemolysis.
* Clinically significant gastrointestinal bleeding or any other clinically significant active bleeding within 3 months prior to study day 1.
* Treatment with another investigational drug or device, or approved therapy for investigational use within 28 days prior to study day 1.
* Pregnancy or lactation for female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ACE-041 in patients with advanced solid tumors or relapsed/refractory multiple myeloma by monitoring adverse events, clinical laboratory tests, vital signs, physical examinations, and anti-drug antibody tests. | 4 months

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic effect of ACE-041 through the collection of blood samples and to evaluate the preliminary anti-tumor activity of ACE-041 through tumor response evaluation, collection of blood biomarkers, and imaging techniques. | 4 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Acceleron Investigative Site, Scottsdale, Arizona
  - Acceleron Investigative Site, Durham, North Carolina
  - Acceleron Investigative Site, Nashville, Tennessee
  - Acceleron Investigative Site, Salt Lake City, Utah